CLINICAL TRIAL: NCT02257684
Title: A Dose Confirmation and Pharmacokinetic Study of Pegcrisantaspase Administered as Intravenous (IV) Infusion in Children and Young Adults With Acute Lymphoblastic Leukemia (ALL) /Lymphoblastic Lymphoma (LBL). Following Hypersensitivity to Pegaspargase (Oncaspar)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-011
Record Dates: First submitted 2014-09-22; First posted 2014-10-06 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: ALL; LBL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegcrisantaspase (Experimental)
  Interventions: Drug: pegcrisantaspase

INTERVENTIONS:
Drug: pegcrisantaspase

SUMMARY:
The purpose of this study is to evaluate the effectiveness,safety, and dosage of pegcrisantaspase in patients with Acute Lymphoblastic Leukemia (ALL) / Lymphoblastic Lymphoma (LBL).

DETAILED DESCRIPTION:
The purpose of the study was to assess the response rate in children and young adults with ALL/LBL and hypersensitivity to pegaspargase defined as the proportion of subjects having a serum asparaginase activity (SAA) level of ≥ 0.1 IU/mL 14 days following the first IV pegcrisantaspase dose in Course 1. Also, to assess the safety of IV pegcrisantaspase therapy in children and young adults with ALL/LBL with hypersensitivity to pegaspargase.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of ALL/LBL
2. Be > 1 to ≤ 21 years of age at study enrollment
3. Have had a ≥ Grade 2 allergic reaction (Common Terminology Criteria for Adverse Events [CTCAE] v4.03) to pegaspargase
4. Have ≥ 1 dose(s) of pegaspargase remaining in his/her treatment plan
5. Have a documented SAA level that is below the limit of quantitation per the analytical method.
6. Subjects must have, in the opinion of the investigator, fully recovered from prior allergic reaction to pegaspargase. Subjects must have completed antihistamine, epinephrine, and/or corticosteroid treatment for the allergic reaction ≥ 24 hours prior to pegcrisantaspase administration.
7. Subjects must have a performance status corresponding to:

   * Karnofsky ≥ 50 (for subjects > 16 years of age)
   * Lansky ≥ 50 (for subjects ≤ 16 years of age)
8. Adequate Renal Function Defined as:

   * Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2 or
   * A serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

   ≥ 16 years 1.7 1.4

   The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR (Schwartz & Gauthier 1985) utilizing child length and stature data published by the CDC.
9. Adequate Liver Function defined as:

   Bilirubin levels ≤ 2.5x ULN for age, and Direct (conjugated) Bilirubin < 0.5 mg/dLSGPT (ALT) ≤ 225 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
10. Subjects who are sexually active must agree to use a medically acceptable method of contraception throughout the entire study period and for 4 weeks after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or the partner include abstinence, birth control pills or patches, diaphragm and spermicide, condom and vaginal spermicide, surgical sterilization, postmenopausal, vasectomy (>6 months prior to baseline), and progestin implant or injection.
11. Able to understand and to sign a written informed consent. All subjects and/or their parent or a legally authorized representative must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Have previously received Erwinia asparaginase
2. Are receiving another investigational agent or will receive an investigational agent in subsequent phases of protocol therapy that include asparaginase
3. Have a history of ≥ Grade 3 pancreatitis (CTCAE v4.03)
4. Prior history of a CNS thrombotic event or ≥ Grade 3 (CTCAE v4.03) thrombotic event, excluding catheter-associated clots
5. Prior history of asparaginase-associated ≥ Grade 3 (CTCAE v4.03) hemorrhagic event or asparaginase-associated thrombus requiring anticoagulation therapy
6. Blood triglyceride levels > 500 mg/dL or > 5.6 mmol/L
7. Hyperglycemia requiring insulin therapy
8. QTc prolongation ≥ 550 msec
9. Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study
10. Subjects who have any serious active disease or co-morbid medical condition (according to investigator's decision), or psychiatric illness that would prevent the subject from signing the informed consent form, assent form or informed consent form by parents, pending institutional requirements, or per investigator's opinion, would prevent the subject from completing one course of pegcrisantaspase.

Pregnant or lactating females or females of childbearing potential not willing to use an adequate method of birth control for the duration of the study. Female subjects who are lactating who do not agree to stop breast-feeding.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skowronski, MD, PhD, Study Director — Jazz Pharmaceuticals
Locations (43):
- United States (43):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital / UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center Center for Cancer & Blood Disorders, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children / Indiana University, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital Main Campus, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - C.S. Mott / University of Michigan, Ann Arbor, Michigan
  - Wayne State University c/o Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Medical Center - Fairview, Minneaplois, Minnesota
  - Children's Hospitals & Clinics of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital & Medical Center of Omaha, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Levine Cancer Institute, Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Bi-Lo Charities Children's Cancer Center, Greenville, South Carolina
  - Vanderbilt University Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital / Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seatlle, Washington
  - University of Wisconsin / American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin / Midwest Children's Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegcrisantaspase: IV administration of pegcrisantaspase in Course 1
Period: Overall Study
Arm/Group | Pegcrisantaspase
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Sponsor's Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Pegcrisantaspase: pegcrisantaspase
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 12.95 [7.8 to 20.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Response Rate in Children & Young Adults With ALL/LBL and Hypersensitivity to Pegaspargase Defined as the Proportion of Subjects Having a Serum Asparaginase Activity (SAA) Level of >= 0.1 IU/mL Following the First IV Dose in Course 1
Time Frame: 15 days during Course 1
Population: Only 1 of the first 4 patients dosed achieved the predefined serum asparaginase activity (SAA) level above the 0.1 IU/mL therapeutic threshold 14 days following the first IV pegcrisantaspase dose in Course 1 (Primary Objective of the study).
Measure: Number; unit: SAA Level IU/mL
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 1
SAA Level IU/mL
  Course 1; Day 0 (Screening) | 0.013
  Course 1; Day 1 (Pre-dose) | 0.013
  Course 1; Day 1 (1 hour post) | 0.50
  Course 1; Day 1 (3 hour post) | 0.44
  Course 1; Day 1 (5 hour post) | 0.41
  Course 1; Day 2 (Visit 2) | 0.36
  Course 1; Day 8 (Visit 3) | 0.28
  Course 1; Day 11 (Visit 4) | 0.24
  Course 1; Day 15 (Visit 5) | 0.26

2. Primary Outcome: The Serum Asparaginase Activity 14 Days After the First Infusion of Study Drug and the Adverse Events in All Participants.
Time Frame: 1 Year
Population: Not Applicable, as the study was terminated before this endpoint was analyzed.
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 0
Value | 0

3. Secondary Outcome: The Pharmakokinetic (PK) Profile of IV Pegcrisantaspase in Children and Young Adults With ALL/LBL and Hypersensitivity to Pegaspargase. Pharmakokinetic Profiles to be Assessed Are: Half Life, Elimination Rate, Tmax, Cmax, AUC.
Time Frame: 14 Days
Population: Not Applicable, as the study was terminated before this endpoint was analyzed.
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 0
Value | 0

4. Secondary Outcome: The SAA Levels Over Time Following Repeated Administration in Children and Young Adults ALL/LBL and Hypersensitivity to Pegaspargase
Time Frame: 30 Days
Population: Not Applicable, as the study was terminated before this endpoint was analyzed.
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 0
Value | 0

5. Secondary Outcome: The Immunogenicity of IV Pegcristaspase by Testing Anti-pegcrisantaspase and Anti-PEG Binding and Neutralizing Antibodies
Time Frame: 30 Days
Population: Not Applicable, as the study was terminated before this endpoint was analyzed.
Arm/Group | Pegcrisantaspase
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | Pegcrisantaspase
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcrisantaspase (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcrisantaspase (N=4)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Periorbital oedema (Eye disorders) | 1
Mucosal inflammation (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Only 1 patient achieved the predefined SAA level above the 0.1 IU/mL therapeutic threshold 14 days following IV pegcrisantaspase dose in Course 1. Therefore, the corresponding PK parameters for repeated administration were not calculated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No